CLINICAL TRIAL: NCT04681989
Title: Moving On Study - Pilot Test
Acronym: MOST-PT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Lynn Sage Breast Cancer Research Foundation (Unknown)
Responsible Party: Principal Investigator, Ann Marie Flores, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STU00206619
Record Dates: First submitted 2020-12-16; First posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Intervention Model Description: Participants were randomized to either the intervention or control group after baseline (within 1 month of completing active, intent-to-cure breast cancer treatment) measurement by research assistants. Follow-up outcome measures at 1 month after baseline.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Biostatistician generated the randomization list. The research assistant called the PI for group assignment after baseline measures were taken.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MOVE-ABC intervention arm (Experimental): MOVE-ABC interventional group participants receive usual care plus the MOVE-ABC education instruction and materials. After the participant completes the baseline assessment (T0) and been given the study survey by a research staff member she will receive the following:
  1. instructions on the education materials by a research staff member
  2. a range of motion wand
  3. a small ball
  4. MOVE-ABC education booklet and video
  The intervention group will complete 4 weekly follow-ups with a research staff member over the phone. The follow-ups will be completed in between the T0 (baseline) assessment, and the T1 (1 month after baseline) assessment. The follow-up phone calls are expected to take 20 - 30 minutes each time. During these follow-ups research staff will review material, and answer any questions the participant may have. All documentation of phone calls and questions asked by participants during these reviews will be captured in REDCap.
  Interventions: Behavioral: Moving On After Breast Cancer
- Control/Usual Care arm (No Intervention): Control group participants will be measured at baseline and at 1 month follow-up. They receive usual care. Usual care does not include specialized, physical therapy-based education on recovery from breast cancer.

INTERVENTIONS:
Behavioral: Moving On After Breast Cancer — After the MOVE-ABC interventional group participant completes their baseline assessment (T0) and been given the study survey by a research staff member she will receive the following:
  1. Instructions on how to use the physical therapy-based education materials by a research staff member
  2. a range of motion wand
  3. a small ball
  4. MOVE-ABC education booklet and video
  The intervention group will complete 4 weekly follow-ups with a research staff member over the phone. The follow-ups will be completed in between the T0 (baseline) assessment, and the T1 (1 month after baseline) assessment.
  Other Names: MOVE-ABC
  Arms: MOVE-ABC intervention arm

SUMMARY:
The purpose of this study is to conduct a pilot test of "Moving On After Breast Cancer (MOVE-ABC)" - a physical therapy based educational intervention designed to reduce and manage breast cancer-related physical and functional impairments. This pilot test will allow the investigator to determine whether MOVE-ABC is feasible and holds promise for efficacy for delivery after breast cancer treatment has ended just as the breast cancer survivor enters the surveillance for recurrence phase of cancer survivorship. The study team will be recruiting breast cancer survivors who have just finished intent-to-cure treatment and are just about to execute their cancer survivorship plans.

DETAILED DESCRIPTION:
The investigators hypothesize that MOVE-ABC is a critical missing link in the standard of care to reduce impairments and improve confidence to manage impairments. The research team is positioned to pilot test MOVE-ABC to address (a) self- management of breast cancer-related impairments via patient-centered booklet and video each impairment identified by our breast cancer survivors; (b) instruction on self-management of impairments with the "Moving On" booklet and video (Attachment 4.1); and (c) weekly follow-up (up to 1 month after the end of breast cancer treatment) to answer questions, concerns and review "Moving On". This research also supports a small but growing number of studies that point to self-management interventions informed by rehabilitation as a means to fill this gap in usual care. The investigator has already piloted the "Moving On" intervention among surgical candidates for breast cancer surgery. The question remains whether "Moving On" is acceptable and feasible for breast cancer survivors who have already completed their breast cancer treatment and are just beginning to execute their breast cancer survivorship plans.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed and treated BC (stages 0-4)
* female
* English speaking
* 21 years old or older

Exclusion Criteria:

* previous history of cancer (except non-melanoma skin)
* history of shoulder impairment (e.g. shoulder osteoarthritis, rotator cuff tear, adhesive capsulitis)
* pregnancy
* central nervous system damage (e.g.: spinal cord injury, brain injury, multiple sclerosis, etc.)
* dementia
* systemic medical conditions and/or metal implants (e.g. fibromyalgia, rheumatoid arthritis, diabetes, joint replacement, cardiac pacemaker, port-a-cath etc.)
* upper extremity(ies) amputation
* actively receiving physical therapy for any reason prior to enrollment

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
EORTC Information-25 (EORTC-QLQ-INFO25) | Change from baseline to 1 month after baseline
  EORTC-QLQ-INFO25 is a 25- item survey with 4 multi-item sub-scales on satisfaction with information on cancer, medical tests, treatment, other services. It has high internal consistency (α>0.90) with sub-scales ranging between .70 -.82. Test-retest reliability is good (intraclass correlation coefficients >0.70). Convergent validity is supported by significant correlation with other information satisfaction surveys (r>0.40).

SECONDARY OUTCOMES:
Self-efficacy for Managing Chronic Disease 6-Item (SEMCD-6) Scale | Change from baseline to 1 month after baseline
  The Self-Efficacy for Managing Chronic Disease 6-Item (SEMCD-6) Scale inquires about self-confidence in prevention of disease side effects (e.g., fatigue, pain, emotional distress, other symptoms) from interfering with daily activity, managing health care needs, and aspects of disease without medication. This scale has been used in cancer and chronic musculoskeletal disease studies.

CONTACTS AND LOCATIONS:
Overall Officials: Ann M Flores, PT, PhD, Principal Investigator — Northwestern University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martins da Silva RC, Rezende LF. Assessment of impact of late postoperative physical functional disabilities on quality of life in breast cancer survivors. Tumori. 2014 Jan-Feb;100(1):87-90. doi: 10.1700/1430.15821. PMID 24675497
- [Background] Binkley JM, Harris SR, Levangie PK, Pearl M, Guglielmino J, Kraus V, Rowden D. Patient perspectives on breast cancer treatment side effects and the prospective surveillance model for physical rehabilitation for women with breast cancer. Cancer. 2012 Apr 15;118(8 Suppl):2207-16. doi: 10.1002/cncr.27469. PMID 22488695
- [Background] Pinto M, Gimigliano F, Tatangelo F, Megna M, Izzo F, Gimigliano R, Iolascon G. Upper limb function and quality of life in breast cancer related lymphedema: a cross-sectional study. Eur J Phys Rehabil Med. 2013 Oct;49(5):665-73. Epub 2013 May 23. PMID 23698473
- [Background] Hack TF, Kwan WB, Thomas-Maclean RL, Towers A, Miedema B, Tilley A, Chateau D. Predictors of arm morbidity following breast cancer surgery. Psychooncology. 2010 Nov;19(11):1205-12. doi: 10.1002/pon.1685. PMID 20099254